CLINICAL TRIAL: NCT05915767
Title: Assessment of Therapeutic Effect of Olive (Olea Europaea L.) Leaf Tea on Gastrointestinal Symptoms and Body Composition in Adults With Small Intestinal Bacterial Overgrowth
Brief Title: Therapeutic Effect of Olive Leaf Tea on SIBO
Acronym: SIBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Sanaullah Iqbal, Professor, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIBO
Record Dates: First submitted 2023-05-18; First posted 2023-06-23 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Small Intestinal Bacterial Overgrowth; Gastrointestinal Disorder, Functional
Keywords: Olive leaf tea; Olive leaf; Body composition; Gastrointestinal symptoms
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two groups. One group will take olive leaf tea, and the other group will receives no tea.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- olive leaf tea (Experimental): SIBO diagnosed individuals in this group will receive olive leaf tea orally, twice a day after meals for 8 weeks.
  Interventions: Dietary Supplement: Olive leaf tea
- Control group (No Intervention): SIBO diagnosed individuals in this group will not receive olive leaf tea or any intervention for 8 weeks.

INTERVENTIONS:
Dietary Supplement: Olive leaf tea — Fresh olive leaves will be procured from Chakwal, Pakistan. The leaves will be rinsed to remove dust and debris and dried at 40℃ in the oven. The leaves will be ground into powder form and then incorporated in tea bags containing 1.8 g leave powder/tea bag. Participants in treatment group will be instructed to dip the tea bag in 200-250 ml boiling water for 3-5 minutes.
  Arms: olive leaf tea

SUMMARY:
The goal of this study is to learn about the effect of olive leaf tea (OLT) in patients with small intestinal bacterial overgrowth aging from 18 to 60 years old. This study aims to answer the following questions:

* Will OLT consumption help decrease severity of gastrointestinal signs and symptoms
* Will OLT help normalize the intestinal methane and hydrogen gases levels measured by glucose breath test
* Does olive leaf tea have an effect on body composition parameters including weight, muscle mass and fat mass Participants with complain of gastrointestinal symptoms like abdominal gas, constipation, diarrhea etc. will undergo glucose breath test(GBT). Participants with diagnosed SIBO by GBT will randomly assigned to two groups. Group A will take the olive leaf tea(1.8g leave powder /tea bag) twice/day after meals for the duration of 2 months. Group B (control group) will not take olive leaf tea. For both groups Symptomatic questionnaire, Glucose breath test, Body composition by InBody analyzer 270 and 24-hour dietary recall will be taken. Researcher will compare readings of group A and Group B taken at Baseline and after 2 months of intervention to assess the effect of Olive leaf tea

DETAILED DESCRIPTION:
Small intestinal bacterial overgrowth (SIBO), characterized by an abnormal increase in the population of overall or harmful bacteria species in the small intestine, resulting in malabsorption, malnutrition, alter body composition and can lead to further complications if not addressed timely. Herbal therapy is considered quite effective in treating SIBO. No literal data is available concerning therapeutic effect of olive leaf tea on SIBO patients. Olive leaves consist of high concentration of phenolic compounds and essential fatty acids that assist in restoring altered gut microbiota and in weight management, also possess significant antimicrobial effect against opportunistic intestinal bacteria. Objective of this study is to evaluate the antimicrobial potential of olive leaf infusion on intestinal microbiota analyzed by hydrogen and methane breath test and its effect on body composition parameters in SIBO individuals. This study will also observe the effect of OLT on gastrointestinal signs and symptoms. This study comprises of 3 phases:

Phase 1: Olive leaf tea preparation

Phase 2: Participants recruitment Study participants will be recruited via circulating SIBO screening questionnaires throughout the university. Individuals with mean symptomatic score (≥4) and fulfilling the inclusion criteria will be examined using a confirmatory test known as the hydrogen/methane breath test (BT). 50g glucose solubilized in 250 mL water given to participants orally. Breath samples will be taken every 15 minutes for 2 hours. After written and oral consent, 50 participants with positive BT results will be included in the study. Experimental design: SIBO-diagnosed individuals will be randomly assigned to two groups (treatment and control) with 25 participants in each group. The treatment group will take tea twice a day after meals for 2 months. Participants will be requested to record the following information daily: consumption of OLT and any side effects if experienced the control group will not receive tea or any other intervention.

Phase 3: Assessment tests: GI symptoms, Hydrogen and methane breath test, 24-hour dietary intake, and body composition analysis will be done before and after the intervention.

Statistical analysis:

Microsoft excel will be used for data coding. Descriptive analysis will be carried out by using SPSS version 23 (SPSS for Windows version 23; SPSS Inc., Chicago, IL, USA). Independent sample t-test and Pearson chi-square test will be used to compare control and treatment groups. Paired sample t-test will be performed to measure within-group differences from the baseline. A chi-square test will be applied to develop a correlation between age, gender, and BMI with SIBO. P<0.05 was considered significant for all analysis

ELIGIBILITY:
Inclusion Criteria:

* positive hydrogen or methane breath test

Exclusion Criteria:

* Hospitalized
* Stroke
* Coronary obstructive pulmonary disease (COPD)
* Cancer
* Diabetes mellitus
* history of GI surgeries except cholecystectomy
* history of GI surgeries except hysterectomy and appendectomy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Gastrointestinal mean symptomatic score at week 8. | Change from baseline mean symptomatic score at 2 months
  Gastrointestinal signs and symptoms will be assessed by using a 9 symptomatic questionnaire for SIBO. It is a validated questionnaire in which individuals will be asked to rate their GI symptoms according to frequency, intensity and duration on a 3 point Likert scale ranging from 0 (no symptom) to 3 (severe symptom).Individuals with a mean score ≥4 will be considered suspect of SIBO.
Normalization of methane and hydrogen levels in breath test | Change from baseline H2 and CH4 levels at 2 months
  Hydrogen and methane level in Breath test will be measured by QuinTron breath tracker SC analyzer. Individuals having ≥12 ppm rise in H2 and/or a ≥10 ppm rise in CH4 from the baseline reading or from the lowest preceding value will be diagnosed as positive for SIBO.

SECONDARY OUTCOMES:
Weight change in kilograms | Change from baseline weight at 2 months
  Electronic weighing scale will be used to assess weight change in both groups.
Change in Body fat mass in kilograms | Change from baseline fat mass at 2 months
  The fat analysis will be done by using InBody 270. It will also tell about percentage of fat in different body segments.
Change in BMI in kg/m^2 | Change from baseline BMI at 2 months
  The BMI will be calculated using weight(kg) and height(m^2).
Change in basal metabolic rate (BMR) in kcal | Change from baseline BMR at 2 months
  The BMR will be calculated using analyzer InBody 270.

CONTACTS AND LOCATIONS:
Overall Officials: Sanaullah Iqbal, PhD, Principal Investigator — University of Veterinary and animal Sciences, Lahore, Punjab, Pakistan.
Locations (1):
- UVAS, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vezza T, Rodriguez-Nogales A, Algieri F, Garrido-Mesa J, Romero M, Sanchez M, Toral M, Martin-Garcia B, Gomez-Caravaca AM, Arraez-Roman D, Segura-Carretero A, Micol V, Garcia F, Utrilla MP, Duarte J, Rodriguez-Cabezas ME, Galvez J. The metabolic and vascular protective effects of olive (Olea europaea L.) leaf extract in diet-induced obesity in mice are related to the amelioration of gut microbiota dysbiosis and to its immunomodulatory properties. Pharmacol Res. 2019 Dec;150:104487. doi: 10.1016/j.phrs.2019.104487. Epub 2019 Oct 11. PMID 31610229
- [Background] Liu Y, McKeever LC, Malik NS. Assessment of the Antimicrobial Activity of Olive Leaf Extract Against Foodborne Bacterial Pathogens. Front Microbiol. 2017 Feb 2;8:113. doi: 10.3389/fmicb.2017.00113. eCollection 2017. PMID 28210244
- [Background] El-Sayed NR, Samir R, Jamil M Abdel-Hafez L, Ramadan MA. Olive Leaf Extract Modulates Quorum Sensing Genes and Biofilm Formation in Multi-Drug Resistant Pseudomonas aeruginosa. Antibiotics (Basel). 2020 Aug 19;9(9):526. doi: 10.3390/antibiotics9090526. PMID 32824901
- [Background] Mujico JR, Baccan GC, Gheorghe A, Diaz LE, Marcos A. Changes in gut microbiota due to supplemented fatty acids in diet-induced obese mice. Br J Nutr. 2013 Aug;110(4):711-20. doi: 10.1017/S0007114512005612. Epub 2013 Jan 10. PMID 23302605
- [Background] Kocyigit A, Guler EM, Irban A, Kiran B, Atayoglu AT. Assessment of Association Between the Potential Immunomodulatory Activity and Drinking Olive Leaf Tea in the Coronavirus Disease-2019 Pandemic: An Observational Study. J Integr Complement Med. 2022 Dec;28(12):940-947. doi: 10.1089/jicm.2022.0554. Epub 2022 Sep 16. PMID 36112183
- [Background] Rocchetti G, Luisa Callegari M, Senizza A, Giuberti G, Ruzzolini J, Romani A, Urciuoli S, Nediani C, Lucini L. Oleuropein from olive leaf extracts and extra-virgin olive oil provides distinctive phenolic profiles and modulation of microbiota in the large intestine. Food Chem. 2022 Jun 30;380:132187. doi: 10.1016/j.foodchem.2022.132187. Epub 2022 Jan 21. PMID 35086016
- [Background] Erdogan A, Rao SS, Gulley D, Jacobs C, Lee YY, Badger C. Small intestinal bacterial overgrowth: duodenal aspiration vs glucose breath test. Neurogastroenterol Motil. 2015 Apr;27(4):481-9. doi: 10.1111/nmo.12516. Epub 2015 Jan 19. PMID 25600077
- [Background] Onana Ndong P, Boutallaka H, Marine-Barjoan E, Ouizeman D, Mroue R, Anty R, Vanbiervliet G, Piche T. Prevalence of small intestinal bacterial overgrowth in irritable bowel syndrome (IBS): Correlating H2 or CH4 production with severity of IBS. JGH Open. 2023 Apr 3;7(4):311-320. doi: 10.1002/jgh3.12899. eCollection 2023 Apr. PMID 37125253
- [Background] Ramirez EM, Brenes M, Romero C, Medina E. Olive Leaf Processing for Infusion Purposes. Foods. 2023 Jan 30;12(3):591. doi: 10.3390/foods12030591. PMID 36766119
- [Background] Sheeza I, Sanaullah Iqbal, Rabbani I, M Asif Ali. 2021. Prevalence of Small Intestinal Bacterial Overgrowth in People with Gastrointestinal Signs and Symptoms Using Glucose Breath Test. Acta Scientific NUTRITIONAL HEALTH (ISSN:2582-1423). 05(12 December 2021).
- [Background] Mattioli LB, Frosini M, Amoroso R, Maccallini C, Chiano E, Aldini R, Urso F, Corazza I, Micucci M, Budriesi R. Olea europea L. Leaves and Hibiscus sabdariffa L. Petals Extracts: Herbal Mix from Cardiovascular Network Target to Gut Motility Dysfunction Application. Nutrients. 2022 Jan 21;14(3):463. doi: 10.3390/nu14030463. PMID 35276825
- [Background] Malfa GA, Di Giacomo C, Cardia L, Sorbara EE, Mannucci C, Calapai G. A standardized extract of Opuntia ficus-indica (L.) Mill and Olea europaea L. improves gastrointestinal discomfort: A double-blinded randomized-controlled study. Phytother Res. 2021 Jul;35(7):3756-3768. doi: 10.1002/ptr.7074. Epub 2021 Mar 16. PMID 33724592
- [Background] Dekaboruah E, Suryavanshi MV, Chettri D, Verma AK. Human microbiome: an academic update on human body site specific surveillance and its possible role. Arch Microbiol. 2020 Oct;202(8):2147-2167. doi: 10.1007/s00203-020-01931-x. Epub 2020 Jun 10. PMID 32524177